CLINICAL TRIAL: NCT06444672
Title: Effects of a Home-Based Rehabilitation on Anthropometric Measures, Sensory-Motor Functions and Independence After Spinal Cord Injury
Acronym: HBRSCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mosul (Other)
Collaborators: University of Sfax (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMosul
Record Dates: First submitted 2024-05-11; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injury at T7-T10 Level; War Injuries Due to Bullets and Fragments; Spinal Cord Injury L1- L5; Spinal Cord Injury No Sensory/Motor in S4-S5
Keywords: Spinal cord Injury; Anthropometric Measures; Muscles Strength; Motor-Sensory Functions; Home-Based Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Serial case study in a quasi-experimental design
Masking Description: Home-based rehabilitation program We used ASIA-scale to evaluate sensory function and voluntary movement7. The HBRP included whole-body training with various exercises for stretching, strength, endurance, and aerobic fitness. The treatment sessions were performed three times per week and had a 50-120-min duration. The exercises were modified based on individual progress and included the use of a rubber ball for balance and strength as well as trunk flexibility, static balance, stability, and standing exercises. Participants who could stand with assistive devices (such as knee-ankle-foot orthoses, KAFO) performed walking exercises.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBRP (Experimental): The HBRP included whole-body training with various exercises for stretching, strength, endurance, and aerobic fitness. The treatment sessions were performed three times per week and had a 50-120-minute duration. The exercises were modified based on individual progress and included the use of a rubber ball for balance and strength as well as trunk flexibility, static balance, stability, and standing exercises.
  Interventions: Other: Home-based Rehabilitation program; Device: Knee-Ankle-Foot-Orthosis

INTERVENTIONS:
Other: Home-based Rehabilitation program — Home-based rehabilitation program The investigators used the ASIA scale to evaluate the sensory function and voluntary movement7. The HBRP included whole-body training with various exercises for stretching, strength, endurance, and aerobic fitness. The treatment sessions were performed three times per week and had a 50-120-minute duration. The exercises were modified based on individual progress and included the use of a rubber ball for balance and strength as well as trunk flexibility, static balance, stability, and standing exercises. Participants who could stand with assistive devices (such as knee-ankle-foot orthoses, KAFO) performed walking exercises.
  Other Names: HBRP
Device: Knee-Ankle-Foot-Orthosis — It is used to assist the participant in holding his /her body weight on the lower limb through standing and walking
  Other Names: KAFO devices

SUMMARY:
Background: The scarcity of resources for spinal cord injury (SCI) rehabilitation constitutes a significant obstacle, particularly in war-torn regions experiencing a rise in such injuries. Implementing a home-based rehabilitative program (HBRP) tailored to patients' environmental, social, and financial contexts is crucial in mitigating this challenge. The authors investigated the effects of a 24-month HBRP on anthropometric measurements, muscular strength, sensory and motor function, and independence in participants transitioning from bed to walking following SCI.

Methods: Serial case study in a quasi-experimental design, the conducting was at the participants' homes. The participants were four patients with SCI (experimental group) and another two patients with SCI (control group). The interventions were a 24-month HBRP comprising strength, flexibility, and balance training, the outcome measures involved anthropometric measurements, muscle strength using a digital handheld dynamometer, muscle thickness, and cross-sectional area measured using magnetic resonance imaging, measured five walking tests, and the American Spinal Injury Association scale (ASIA) score for assess the sensory and motor score, and the Spinal Cord Independence Measure (SCIM).

DETAILED DESCRIPTION:
Materials and Methods

The primary condition being studied:

Spinal Cord Injury Paraplegia according to ASIA-scale Type A Complete damage No Sensory/Motor in S4-5

Participants

From (NRCODP), the authors accessed six participants with SCIs who participated voluntarily in this study (three males and one female; their mean age was 24.75 years). Those patients constituted the experimental group. Their injuries were classified as grade A according to the American Spinal Injury Association (ASIA) scale. Spinal cord damage was observed at T6, T8, L1, and L2. The participants started receiving the HBRP intervention 4-6 months after injury and the program lasted 24 months. The control group comprised two volunteers (mean age 23.50 years) with SCIs at T9 and L1. These patients only served as a comparison for magnetic resonance imaging (MRI) findings.

This study was a case series that included a home-based therapeutic exercise program. Strength and ASIA- scales were assessed every 6 months. The walking evaluation was performed monthly for 10 months after the participants began using assistive devices. The final assessment was conducted at 24 months.

Home-based rehabilitation program The investigators used the ASIA scale to evaluate sensory function and voluntary movement. The HBRP included whole-body training with various exercises for stretching, strength, endurance, and aerobic fitness. The treatment sessions were performed three times per week and had a 50-120-minute duration. The exercises were modified based on individual progress and included using a rubber ball for balance and strength, as well as trunk flexibility, static balance, stability, and standing exercises. Participants who could stand with assistive devices such as knee-ankle-foot orthoses (KAFO) performed walking exercises. During the 24 months, the program encountered technical obstacles during implementation, primarily related to the unavailability of suitable tools to optimize exercise performance while ensuring participant safety, especially during the first 6 months. Precautionary measures included creating a secure exercise environment within a furniture-free 2-meter square, employing safety belts, maintaining a safe distance, and involving participants' relatives for assistance, especially during the introduction of new and challenging motor tasks. Participants' families either purchased or received exercise equipment, and some devices were locally manufactured based on standard specifications. Participants facing negative psychological states due to motor challenges and monotony received psychological, faith-based, encouraging, and entertaining interventions, incorporating real-life success stories through video observations of individuals with SCIs. During the 24 months, the program encountered technical obstacles during implementation, primarily related to the unavailability of suitable tools to optimize exercise performance while ensuring participant safety, especially during the first 6 months. However, precautionary measures included creating a secure exercise environment within a furniture-free 2-meter square, employing safety belts, maintaining a safe distance, and involving participants' relatives for assistance, especially during the introduction of new and challenging motor tasks. Participants' families either purchased or received exercise equipment, and some devices were locally manufactured based on standard specifications. Participants facing negative psychological states due to motor challenges and monotony received psychological, faith-based, encouraging, and entertaining interventions, incorporating real-life success stories through video observations of individuals with SCIs.

Walking tests. The 10-m walk test (WT), 2-min WT (2MWT), 4MWT, 6MWT, and Up & GO (WT) were used when the participants reached the walking phase. These tests were used to assess walking speed improvement and endurance in patients with SCI. The investigators chose wide, suitable areas at participants' homes for walking assessments to adhere to test prerequisites. Essential equipment, including markers denoting starting and concluding points, was supplied and distinguished "Remember the following text: 'by colorful stickers'", stopwatches, and measuring tapes. Further, safety protocols were implemented to safeguard participants during test execution, and all tests were carried out according to the relevant standards.

In addition, a kinesthetic analysis approach was used, in which mental visualization played a pivotal role in patients who lack a sense of balance. Locally manufactured assistive devices (e.g., KAFO) were used, and coordination between doctors and the author ensured effective treatment and successful rehabilitation.

Outcome measures Anthropometric measurements, including the abdominal, pelvic, thigh, and leg circumference, were taken using a tape measure. Weight and height were measured using traditional scales. Patient measurements (weight, body mass index [BMI], and anthropometric measurements) were monitored every 6 months throughout the intervention period. The ASIA scale was used to examine the sensory and motor function before stating HBRP and subsequently every 6 months. The pre-HRBP and 24-month values were also compared. In addition, muscle strength was measured using a Micro-FET2 dynamometer (Hoggan Scientific LLC, Salt Lake City, UT), where the participants exerted maximum force against the device while the examiner provided resistance. The tests lasted a few seconds and were signalled by the commands "go" and "relax". The Spinal Cord Independence Measure (SCIM) includes the self-care (0-20), respiration and sphincter management (0-40), and mobility (0-40) sub-scores. Each area is scored according to its proportional weight in these patients' general activity. The final score ranges from 0 to 100, with a high score indicating higher independence, the authors assess the independence of participants during the 24 months of rehabilitation.

Magnetic resonance imaging technical considerations MRI examinations were performed in the supine position using a hybrid 1.5 T MRI scanner (Elekta Unity™, Philips, Stockholm, Sweden), which is a modified 1.5 T Philips Ingenia (Best, The Netherlands). Long stair and T1 fat suppression sequences were used to investigate the utility of MRI in measuring changes in muscle volume, and anatomical cross-sectional area (CSA), focusing on the rectus femoris (RF) and gluteus maximus (GM) muscles. Additionally, the MRIs included muscle thickness (MT) in (mm) and CSA measurements for the bilateral RF and GM muscles. These measurements were repeated 8-9 months after the start of standing and walking training. Previous research has already established the reliability and validity of MRI for measuring MT and its capability to detect and monitor muscle changes during immobilization.

During MRI analysis, the initial peak corresponds to muscle density, while the subsequent peak indicates fat density, and the midpoint between these peaks delineates muscle from fat pixels. Calculations of CSAs were performed using the equations outlined by Gorge and Dudley. Muscle CSA (cm2) = ¼ of the total number of muscle pixels * ([field of view {FOV} / matrix size])2, and Intramuscular Fat (IMF) CSA (cm2) = ¼ of the total number of IMF pixels * ([FOV / matrix size])2. To normalize for skeletal muscle size discrepancies across groups, IMF CSA was expressed relative to skeletal muscle CSA: Relative IMF = ¼ of ([IMF CSA / muscle CSA] * 100).

Statistical analysis Study outcomes were compared across time points using a one-way repeated-measures analysis of variance. The ES was quantified by Cohen's criteria. Additionally, paired sample t-tests were used to compare pre-and post-intervention MRI measures and ASIA scale scores. SPSS version 24.0 (IBM Corp., Armonk, NY, USA) was used for all analyses. An alpha value <0.05 indicated statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Every patient has SCI resulting from the ISIS war and HE/SHE committed to implementing the HBRP without interruption and implements all instructions from the researcher supervising the program.

Exclusion Criteria:

* If any information and conditions above are not available.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements | Every 6-month repeated measures follow-up for 24 months
  The abdominal, pelvic, thigh, and leg circumferences were taken using a tape measure depending on the centimeter (cm) unit from the lying down position. These measures were measured to determine the changes in morphological shape for those parts as a result of home-based rehabilitation for 24 months. This was done using repeated measures that included multiple axes, in addition to others, such as muscle strength. Certain anthropometric measurements, quantified in centimeters, were chosen to monitor alterations arising from the efficacy of the Home-Based Rehabilitation Program (HBRP). These selected measurements comprised Waist/Abdomen circumference, Pelvis circumference, Right/Left Thigh circumference, and Right/Left Leg circumference. Anthropometric parameters, encompassing the circumference of various body segments, were diligently documented through the application of a tape measure.
Weight, height, and body mass index BMI | Every 6-month and follow-up for 24 months
  Encompassed weight and body mass index (BMI) was consistently tracked, with specific consideration given to injury-related factors. The height was measured in (cm), and the weight was measured by using traditional scales in (kg). Both weight and height were used to measure the body mass index (BMI). These measures were repeated every 6 months for 24 months to follow up the changes in body weight according to increasing the activity and metabolic in muscles after a home-based rehabilitation program (HBRP).
The American Spinal Injury Association ( ASIA) scale | Every 6-month and follow-up for 24 months
  It was used to examine the sensory and motor function before and after starting a home-based rehabilitation program (HBRP). The clinical evaluation incorporated the application of the American Spinal Injury Association ( ASIA) scale to measure sensory perception and the potential for voluntary movement, the degree from (0-100) as following the guidelines. Furthermore, the ASIA scale was employed in alignment with an interval of HBRP to appraise participants' sensory and motor function levels to assess the effectiveness of the rehabilitation program, drawing parallels with the methodology utilized. Additionally, ASIA was executed to gauge sensory perception and the capacity for voluntary movement on both sides of the participants' bodies, following the framework outlined.
Muscle strength | Every 6-month and follow-up for 24 months
  It involved the lower extremity, head, trunk, and pelvis muscle strength tests as a result of HBRP. Muscular strength was assessed in kilograms (kg) for muscles implicated in lower limb activities below the spinal lesion level, muscular strength was appraised for muscles linked to the Head, Trunk, and Pelvis, operating below the level of the spinal lesion. Utilizing the Micro-FET2 dynamometer by HOGGAN, participants exerted maximal force against the device while the examiner applied resistance to gauge muscle strength. These assessments are initiated through verbal commands ("Go" and "Relax").
  Precautionary measures included creating a secure exercise environment within a furniture-free 2-meter square, employing safety belts, maintaining a safe distance, and involving participants' relatives for assistance, especially during the introduction of new and challenging motor tasks.
Spinal Cord Independence Measure (SCIM) | Every 6-month repeated measures follow-up for 24 months
  The final score ranges from 0 to 100, with a high score indicating a higher independence. A scale was used to assess the level of independence during the 24 months of rehabilitation. This scale involves several items. Its scoring system is self-explanatory; therefore there isn't a manual to instruct the clinician in the scoring process. Scores range from 0-100, where a score of 0 defines total dependence and a score of 100 is indicative of complete independence. Each subscale score is evaluated within the 100-point scale (self-care: 0-20; respiration and sphincter management: 0-40; mobility.
Magnetic resonance imaging (MRI) | 8-9 months after the start of standing and walking training
  MRI examinations were performed in the supine position using a hybrid 1.5 T MRI scanner, which is a modified 1.5 T Philips Ingenia. Long stair and T1 fat suppression sequences were used to investigate the utility of MRI in measuring changes in muscle volume, and anatomical cross-sectional area (CSA) (mm2), focusing on the rectus femoris (RF) and gluteus maximus (GM) muscles. Additionally, the MRIs included muscle thickness (MT) in (mm) and CSA measurements for the bilateral RF and GM muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Munib A Fathe, PhD, Study Chair — University of Mosul
Locations (1):
- Munib Abdullah Fathe, Duhok, Iraq

IPD SHARING:
Plan to Share IPD: Yes
After we complete the publication of this study, we will declare that our data and program will be available by request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication one month
Access Criteria: It should be academically study which hold the same interest

REFERENCES:
- [Background] Akita S, Tokumoto H, Yamaji Y, Ishigaki T, Ogata H, Tezuka T, Kosaka K, Kuriyama M, Mitsukawa N. Comparison of Vectra three-dimensional stereophotogrammetry measurement and tape measurement in the evaluation of perioperative volume change of the lower abdomen in association with lymphatic microsurgery. Microsurgery. 2022 Jan;42(1):50-56. doi: 10.1002/micr.30688. Epub 2020 Nov 23. PMID 33230882
- [Background] Willi R, Widmer M, Merz N, Bastiaenen CHG, Zorner B, Bolliger M. Validity and reliability of the 2-minute walk test in individuals with spinal cord injury. Spinal Cord. 2023 Jan;61(1):15-21. doi: 10.1038/s41393-022-00847-1. Epub 2022 Aug 23. PMID 35999254
- [Background] Kirshblum S, Botticello A, Benedetto J, Donovan J, Marino R, Hsieh S, Wagaman N. A Comparison of Diagnostic Stability of the ASIA Impairment Scale Versus Frankel Classification Systems for Traumatic Spinal Cord Injury. Arch Phys Med Rehabil. 2020 Sep;101(9):1556-1562. doi: 10.1016/j.apmr.2020.05.016. Epub 2020 Jun 10. PMID 32531222
- [Background] Dubinski D, Kolesnyk V. War in Ukraine: a neurosurgical perspective. Acta Neurochir (Wien). 2022 Dec;164(12):3071-3074. doi: 10.1007/s00701-022-05388-3. Epub 2022 Oct 20. PMID 36264367
- [Background] 1. Jesus TS, Landry MD, Hoenig H, Kamenov K, Mills JA, Chatterji S, et al. Global need for physical rehabilitation: Systematic analysis from the global burden of disease study 2019. Lancet. 2020;396:2006-17. doi:10.1016/S0140-6736(20)32340-0
- [Result] Roberts TT, Leonard GR, Cepela DJ. Classifications In Brief: American Spinal Injury Association (ASIA) Impairment Scale. Clin Orthop Relat Res. 2017 May;475(5):1499-1504. doi: 10.1007/s11999-016-5133-4. Epub 2016 Nov 4. No abstract available. PMID 27815685
- [Result] Mohr T, Andersen JL, Biering-Sorensen F, Galbo H, Bangsbo J, Wagner A, Kjaer M. Long-term adaptation to electrically induced cycle training in severe spinal cord injured individuals. Spinal Cord. 1997 Jan;35(1):1-16. doi: 10.1038/sj.sc.3100343. PMID 9025213
- [Result] Frey VN, Renz N, Thomschewski A, Langthaler PB, Schalkwijk FJ Van, Trinka E, et al. applied sciences Influence of Sports on Cortical Connectivity in Patients with Spinal Cord Injury-A High-Density EEG Study. Appl Sci. 2023;13:9469. doi:10.3390/app13169469.
- [Result] Waters RL, Yakura JS, Adkins RH, Sie I. Recovery following complete paraplegia. Arch Phys Med Rehabil. 1992 Sep;73(9):784-9. PMID 1514883
- [Result] Rahimi M, Torkaman G, Ghabaee M, Ghasem-Zadeh A. Advanced weight-bearing mat exercises combined with functional electrical stimulation to improve the ability of wheelchair-dependent people with spinal cord injury to transfer and attain independence in activities of daily living: a randomized controlled trial. Spinal Cord. 2020 Jan;58(1):78-85. doi: 10.1038/s41393-019-0328-7. Epub 2019 Jul 16. PMID 31312016
- [Result] Taccola G, Sayenko D, Gad P, Gerasimenko Y, Edgerton VR. And yet it moves: Recovery of volitional control after spinal cord injury. Prog Neurobiol. 2018 Jan;160:64-81. doi: 10.1016/j.pneurobio.2017.10.004. Epub 2017 Nov 2. PMID 29102670
- [Result] Spungen AM, Asselin PK, Fineberg DB, Kornfeld SD, Harel NY. Exoskeletal-Assisted Walking for Persons with Motor-Complete Paraplegia. New York (NY): VA Rehabilitation Research and Development National Center of Excellence for the Medical Consequences of Spinal Cord Injury. 2013;Feb 4;1-14. [accessed]. http://www.ryzur.com.cn/uploadfile/2016/0830/20160830115519272.pdf
- [Result] Yang A, Asselin P, Knezevic S, Kornfeld S, Spungen AM. Assessment of In-Hospital Walking Velocity and Level of Assistance in a Powered Exoskeleton in Persons with Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):100-9. doi: 10.1310/sci2102-100. Epub 2015 Apr 12. PMID 26364279
- [Result] Mehrholz J, Kugler J, Pohl M. Locomotor training for walking after spinal cord injury. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD006676. doi: 10.1002/14651858.CD006676.pub3. PMID 23152239
- [Result] Richard-Denis A, Dionne A, Mputu PM, Mac-Thiong JM. Do all patients with functional motor-incomplete (AIS-D) traumatic spinal cord injury need specialized inpatient functional rehabilitation? A prospective observational cohort study proposing clinical criteria for home-based rehabilitation after acute care. J Spinal Cord Med. 2024 Sep;47(5):753-764. doi: 10.1080/10790268.2023.2200354. Epub 2023 Apr 21. PMID 37083554
- [Result] van Duijnhoven E, Koopman FS, Ploeger HE, Nollet F, Brehm MA. Effects of specialist care lower limb orthoses on personal goal attainment and walking ability in adults with neuromuscular disorders. PLoS One. 2023 Jan 18;18(1):e0279292. doi: 10.1371/journal.pone.0279292. eCollection 2023. PMID 36652463
- [Result] McIntosh K, Charbonneau R, Bensaada Y, Bhatiya U, Ho C. The Safety and Feasibility of Exoskeletal-Assisted Walking in Acute Rehabilitation After Spinal Cord Injury. Arch Phys Med Rehabil. 2020 Jan;101(1):113-120. doi: 10.1016/j.apmr.2019.09.005. Epub 2019 Sep 27. PMID 31568761
- [Result] Rankin KC, O'Brien LC, Gorgey AS. Quantification of trunk and android lean mass using dual energy x-ray absorptiometry compared to magnetic resonance imaging after spinal cord injury. J Spinal Cord Med. 2019 Jul;42(4):508-516. doi: 10.1080/10790268.2018.1438879. Epub 2018 Feb 20. PMID 29461936
- [Result] Gorgey AS, Shepherd C. Skeletal muscle hypertrophy and decreased intramuscular fat after unilateral resistance training in spinal cord injury: case report. J Spinal Cord Med. 2010;33(1):90-5. doi: 10.1080/10790268.2010.11689681. PMID 20397451